CLINICAL TRIAL: NCT03411421
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Repeated Dosing Regimens of AL-794 in Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Repeated Dosing Regimens of AL-794 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed as the data received to date did not support continuation of the study.
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AL-794-806; AL-794-806 (Other: Alios Biopharma Inc.); 2017-004193-34 (EudraCT Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — sfericase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (AL-794 or Placebo) (Experimental): Participants will receive AL-794 or placebo in 2:1 ratio in Cohorts 1 to 3. AL-794 will be administered at a 100 milligram (mg) loading dose (LD) on the morning of Day 1, followed by a 50 mg maintenance dose (MD) on the evening of Day 1 and twice-daily (BID) on Day 2 through Day 5. The duration of dosing may be extended (maximum duration 10 days), at the discretion of the Sponsor and Principal Investigator (PI).
  Interventions: Drug: AL-794; Drug: Placebo
- Part 2 (AL-794 or Placebo) (Experimental): Participants will receive AL-794 or placebo in 2:1 ratio. AL-794 will be administered as 100 mg LD on the morning of Day 1, followed by a 50 mg MD on the evening of Day 1 and BID on Day 2 through Day 5. The duration of dosing may be extended (maximum duration 10 days). Based on the results of Part 1, the duration of dosing may be modified.
  Interventions: Drug: AL-794; Drug: Placebo

INTERVENTIONS:
Drug: AL-794 — AL-794 will be administered as tablets orally on Day 1 to Day 5.
Drug: Placebo — Matching placebo tablets will be administered.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability (including incidence of central nervous system [CNS] related events such as lightheadedness and dizziness), of multiple oral doses of AL-794 in healthy volunteers (HV). Also, to evaluate the pharmacokinetics of ALS-033719 and ALS-033927 in plasma after multiple oral doses of AL-794 in HV.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written informed consent
* In the Investigator's opinion, the participant is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned
* Participant is deemed healthy on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening
* Body mass index (BMI) 18 - 32 kilogram per meter square (kg/m^2), inclusive. The minimum weight is 50 kilogram (kg). No more than 25 percent (%) of participants may be enrolled with a BMI greater than or equal to (>=) 30 kg/m^2
* Female participants must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening and on Day -1 (admission)

Exclusion Criteria:

* Female who is pregnant as confirmed by a positive beta-human chorionic gonadotropin (beta-hCG) laboratory test, or who was pregnant within 6 months prior to study start, or who is breast-feeding, or who is planning to become pregnant from signing of the informed consent form (ICF) until 90 days after the last dose of study drug
* Male whose female partner is pregnant or contemplating pregnancy from the date of screening until 90 days after their last dose of study drug
* Participant with one or more of the following laboratory abnormalities at screening: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >= 1.2*upper limit of normal (ULN); Alkaline phosphatase (ALP) >= 1.2*ULN; Total bilirubin >= 1.2*ULN; Clinically significant laboratory abnormalities or abnormalities which are deemed to interfere with the ability to interpret study data
* Creatinine clearance less than (<) 90 milliliter per minute (mL/min) (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
* Positive screening test for human immunodeficiency virus type 1 (HIV-1) or HIV-2 antibody, or for current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen [HBsAg]), or hepatitis C virus (HCV) infection (confirmed by HCV antibody) at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 40 days
  An AE is any untoward medical occurrence in a participant who received study drug or placebo without regard to possibility of causal relationship.
Part 1: ALS-033719 Plasma Concentrations | Predose up to Day 12
  Plasma concentration assessment will be done for ALS-033719 following multiple doses of AL-794.
Part 2: ALS-033719 Plasma Concentrations | Predose up to Day 5
  Plasma concentration assessment will be done for ALS-033719 following multiple doses of AL-794.
Part 1: ALS-033927 Plasma Concentrations | Predose up to Day 12
  Plasma concentration assessment will be done for ALS-033927 following multiple doses of AL-794.
Part 2: ALS-033927 Plasma Concentrations | Predose up to Day 5
  Plasma concentration assessment will be done for ALS-033927 following multiple doses of AL-794.

SECONDARY OUTCOMES:
Part 1: ALS-033719 Plasma Concentrations in Healthy Women in Fasted and Fed Conditions | Predose up to Day 12
  Plasma concentration assessment will be done for ALS-033719, after repeated oral doses of AL-794, in healthy women under fasted and fed conditions.
Part 1: ALS-033927 Plasma Concentrations in Healthy Women in Fasted and Fed Conditions | Predose up to Day 12
  Plasma concentration assessment will be done for ALS-033927, after repeated oral doses of AL-794, in healthy women under fasted and fed conditions.
Part 1 and Part 2: Time-Matched Q-T Interval Corrected for Heart Rate Using Fridericia Method (QTcF) | Up to 40 days
  The QTcF will be measured by electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, MD, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom